CLINICAL TRIAL: NCT02458534
Title: The Comparison of Mcgrath Mac, C-MAC, and Macintosh Laryngoscope in Novice Users: a Manikin Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1-2015-0020
Record Dates: First submitted 2015-05-26; First posted 2015-06-01 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: Simulated manikin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mcgrath Mac videolaryngoscope (Experimental): Participants perform three intubation attempts using Mcgrath Mac videolaryngoscope in the manikin with the normal airway setting. Then the participants perform three intubation attempts using the manikin with difficult airway setting.
  Interventions: Other: Mcgrath Mac videolaryngoscope
- C-MAC videolaryngoscope (Experimental): Participants perform three intubation attempts using C-MAC videolaryngoscope in the manikin with the normal airway setting. Then the participants perform three intubation attempts using the manikin with difficult airway setting.
  Interventions: Other: C-MAC videolaryngoscope
- Macintosh laryngoscope (Active Comparator): Participants perform three intubation attempts using macintosh laryngoscope in the manikin with the normal airway setting. Then the participants perform three intubation attempts using the manikin with difficult airway setting.
  Interventions: Other: macintosh laryngoscope

INTERVENTIONS:
Other: Mcgrath Mac videolaryngoscope — Participants perform three intubation attempts using Mcgrath Mac videolaryngoscope in the manikin with the normal airway and difficult airway settings.
  Arms: Mcgrath Mac videolaryngoscope
Other: C-MAC videolaryngoscope — Participants perform three intubation attempts using C-MAC videolaryngoscope in the manikin with the normal airway and difficult airway settings.
  Arms: C-MAC videolaryngoscope
Other: macintosh laryngoscope — Participants perform three intubation attempts using macintosh laryngoscope in the manikin with the normal airway and difficult airway settings.
  Arms: Macintosh laryngoscope

SUMMARY:
The purpose of this study is to evaluate whether the McGrath MAC videolaryngoscope is superior when compared to the C-MAC videolaryngoscope and the Macintosh laryngoscope for novice users in manikin.

ELIGIBILITY:
Inclusion Criteria:

* Medical students

Exclusion Criteria:

* wrist disease excluded.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
time to intubation | within 3 minutes after the insertion of the laryngoscope into the mouth of the manikin
  Time to intubation is defined as the time from the insertion of the laryngoscope into the mouth of the manikin to the confirmation of the chest movement of the manikin.

SECONDARY OUTCOMES:
success rate of the first intubation attempt | Within 3 minutes after the insertion of the laryngoscope into the mouth of the manikin